CLINICAL TRIAL: NCT04737096
Title: DAOIB Combined With tDCS for Early-phase Dementia - a Randomized, Double-blinded and Placebo Controlled Clinical Trial
Brief Title: DAOIB Combined With tDCS for Early-phase Dementia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 201601789A0C603
Record Dates: First submitted 2021-01-27; First posted 2021-02-03 (Actual); Last update posted 2023-01-06 (Actual); Status verified 2023-01

CONDITIONS: Transcranial Direct Current Stimulation; Dementia
MeSH Terms: conditions — Dementia | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tDCS+DAOIB (Experimental)
  Interventions: Drug: DAOIB; Device: tDCS
- tDCS+placebo (Placebo Comparator)
  Interventions: Drug: Placebo; Device: tDCS

INTERVENTIONS:
Drug: DAOIB — The DAOIB dose will be adjusted every 8 weeks according to clinical evaluation.
  Arms: tDCS+DAOIB
Drug: Placebo — placebo
  Arms: tDCS+placebo
Device: tDCS — tDCS

SUMMARY:
This is a 24-week randomized, double-blind, placebo-controlled trial. We will enroll patients with aMCI or mild AD. All patients will receive 2 weeks of tDCS (5 sessions per week, 10 sessions in total) during the first 2 weeks of the study, and will also be allocated randomly to either of 2 treatment groups for 24 weeks: (1) DAOIB group; (2) placebo group. We will assess the patients every 8 weeks during the treatment period (weeks 0, 8, 16, and 24). We hypothesize that augmentation with DAOIB will yield better effect than tDCS alone in improving the cognitive function, global functioning and quality of life in patients with aMCI or mild AD.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Alzheimer's disease or mild cognitive impairment
* MMSE between 10-26
* CDR 1 or 0.5

Exclusion Criteria:

* Hachinski Ischemic Score > 4
* Substance abuse/dependence
* Parkinson disease, epilepsy, dementia with psychotic features
* Major depressive disorder
* Major physical illnesses
* Severe visual or hearing impairment

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-01-02 (Actual); Study Completion 2023-01-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the Alzheimer's disease assessment scale - cognitive subscale at week 8, 16 and 24 | week 0, 8, 16, 24
  Alzheimer's disease assessment scale-cognitive subscale scores range from 0 (best) to 70 (worst)

SECONDARY OUTCOMES:
Change from baseline in Clinician's Interview-Based Impression of Change plus Caregiver Input score at week 8, 16 and 24 | week 8, 16, 24
  Change from baseline in Clinician's Interview-Based Impression of Change plus Caregiver Input score at week 8, 16 and 24
Change from baseline in Mini-Mental Status examination score at week 8, 16 and 24 | week 0, 8, 16, 24
  Change from baseline in Mini-Mental Status examination score at week 8, 16 and 24
Change from baseline in Alzheimer's disease Cooperative Study scale for ADL in MCI (ADCS-MCI-ADL) score at week 8, 16 and 24 | week 0, 8, 16, 24
  The assessment appears to be a suitable instrument for evaluating activities of daily living in early-phase dementia. Its scores range from 0 (worst) to 78 (best)
Change from baseline in Quality of life score at week 8, 16 and 24 | week 0, 8, 16, 24
  Quality of life will be assessed by Medical Outcomes Study Short-Form-36 (SF-36). The SF-36 consists of eight sections: (1) vitality, (2) physical functioning, (3) bodily pain, (4) general health perceptions, (5) physical role functioning, (6) emotional role functioning, (7) social role functioning, and (8) mental health.
Change from baseline in the composite score of a battery of additional cognitive tests at week 24 | week 0, 24
  The battery of additional cognitive tests include speed of processing (Category Fluency), working memory (Wechsler Memory Scale, Spatial Span), verbal/nonverbal learning and memory tests (Wechsler Memory Scale, Word Listing)

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No